CLINICAL TRIAL: NCT00386035
Title: HIV Transmission Risk Behavior Substudy
Brief Title: Effects of Two Anti-HIV Drug Regimens on HIV Transmission Risk Behavior Among SMART Study Participants
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Community Programs for Clinical Research on AIDS (Network)
Responsible Party: Sponsor
Other Study IDs: CPCRA 065B; SMART; 10113 (Registry Identifier: DAIDS-ES)
Record Dates: First submitted 2006-10-06; First posted 2006-10-11 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Treatment Experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: DC Group: HIV infected participants who will stop or defer ART until the CD4 cell count drops below 250 cells/mm3 and who discontinue ART when CD4 cell count reaches above 350 cells/mm3. Participants are followed by episodic ART based on CD4 cell count.
  Interventions: Drug: Delayed ART
- 2: VS Group: HIV infected participants who continue ART to keep viral loads as low as possible, regardless of CD4 cell count.
  Interventions: Drug: Continuous ART

INTERVENTIONS:
Drug: Delayed ART — Participants follow a drug conservation (DC) regimen in which ART is stopped or deferred until CD4 cell count dropped below 250 cells/mm3, initiated until CD4 cell count is at least 350 cells/mm3, and then are followed by episodic ART based on CD4 cell count.
  Groups: 1: DC Group
Drug: Continuous ART — Group 2 participants follow a viral suppression (VS) regimen in which ART was continued to keep viral loads as low as possible, regardless of CD4 cell count.
  Groups: 2: VS Group

SUMMARY:
The purpose of this study is to compare the effects of two different anti-HIV drug regimens on HIV transmission risk behavior among SMART study participants.

DETAILED DESCRIPTION:
It is important to consider the role that HIV infected individuals play in ongoing HIV transmission. Different anti-HIV treatment regimens may lead to variations in HIV transmission risk behavior among HIV infected individuals. HIV infected people with viral loads of less than 1,000 copies/ml are less likely to transmit HIV through heterosexual sex. However, condom use sometimes decreases after individuals start combination antiretroviral therapy (ART); also, some studies have shown an increased rate in acquiring sexually transmitted infections (STIs) following initiation of ART, and those on ART may transmit a drug-resistant strain of HIV. In the SMART study, participants were randomly assigned to one of two treatment groups:

* Group 1 participants will follow a drug conservation (DC) regimen in which ART will be stopped or deferred until CD4 cell count drops below 250 cells/mm3, will be initiated until CD4 cell count is at least 350 cells/mm3, and then will be followed by episodic ART based on CD4 cell count.
* Group 2 participants will follow a viral suppression (VS) regimen in which ART is continued to keep viral loads as low as possible, regardless of CD4 cell count.

The purpose of this study is to compare how the DC and VS regimens affect HIV transmission risk behavior among SMART study participants.

At baseline, participants will complete a questionnaire about their sexual behavior during the previous 2 months. They will also undergo urine and blood collection for STI testing. These same procedures will occur at Months 4 and 12, then every year thereafter for the first 4 years that a participant is in the parent study. Participants and their physicians will be notified of STI testing results so that patients can be referred to appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Coenrollment in the SMART study
* Parent or guardian willing to provide informed consent, if applicable

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV infected participants with a CD4+ cell count greater than 350 cells/mm3 currently receiving or not receiving ART.
Sampling Method: Non-Probability Sample
Enrollment: 883 (Actual)
Dates: Start 2002-01; Primary Completion 2006-01 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To compare the DC group to the VS group for HIV transmission and risk behaviors | At the end of study

SECONDARY OUTCOMES:
To compare the VS group to the DC group on HIV transmission risk behavior in participants who are not on ART at enrollment | At the end of study
To compare the effects of continuing ART in the VS group to stopping ART in the DC group on HIV transmission risk behavior among participants who are on ART at enrollment | At the end of study
To evaluate the correlation between self-reported adherence to ART and HIV transmission risk behavior for participants on ART | At the end of study
To compare the DC and VS groups for HIV transmission risk behavior in subgroups defined by age, gender, possible transmission category, HIV RNA level, and baseline genotypic resistance pattern. | At the end of study
To evaluate the correlation between self-reported transmission risk behavior and the acquisition of certain sexually transmitted diseases as specified in the protocol. | At the end of study
To develop analytic techniques to combine behavioral and biological data into a measure of overall transmission risk | At the end of study

CONTACTS AND LOCATIONS:
Overall Officials: Wafaa El-Sadr, MD, MPH, Study Chair — Harlem AIDS Treatment Group, Harlem Hospital Center; James Neaton, PhD, Study Chair — CPCRA Statistical and Data Management Center/CCBR
Locations (58):
- United States (58):
  - AIDS Healthcare Foundation CRS, Beverly Hills, California
  - UCSF, Fresno, School of Medicine, Dept. of Internal Medicine CRS, Fresno, California
  - Dr. M. Estes Med. Practice CRS, Mill Valley, California
  - Dr. Robert Scott Med. Practice CRS, Oakland, California
  - East Bay AIDS Ctr. CRS, Oakland, California
  - Dr. Shawn Hassler Med. Practice CRS, San Francisco, California
  - Positive Health Program Clinic (San Francisco Gen. Hosp.) CRS, San Francisco, California
  - Dr. Virginia Cafaro Med. Practice CRS, San Francisco, California
  - Dr. William Owen Med. Practice CRS, San Francisco, California
  - Castro-Mission Health Ctr. CRS, San Francisco, California
  - San Francisco VAMC, Infectious Diseases Clinic CRS, San Francisco, California
  - UCSF PHP, Gen. Internal Medicine Practice CRS, San Francisco, California
  - Beacon Clinic at Boulder CRS, Boulder, Colorado
  - Denver Infectious Diseases Consultants CRS, Denver, Colorado
  - Kaiser Permanente of Denver CRS, Denver, Colorado
  - Univ. of Colorado Health Science Ctr. CRS, Denver, Colorado
  - Denver Public Health CRS - INSIGHT, Denver, Colorado
  - Denver Public Health CRS, Denver, Colorado
  - Eastside Family Health Ctr. CRS, Denver, Colorado
  - Denver VAMC CRS, Denver, Colorado
  - Western Infectious Disease Consultants CRS, Wheat Ridge, Colorado
  - Washington DC VAMC, Washington Regional AIDS Program, Infectious Diseases CRS, Washington D.C., District of Columbia
  - Miami VAMC CRS, Miami, Florida
  - Atlanta VAMC CRS, Decatur, Georgia
  - Harper Hosp., Detroit CRS, Detroit, Michigan
  - Wayne State Univ. CRS, Detroit, Michigan
  - Wayne State Univ. INSIGHT CRS, Detroit, Michigan
  - Detroit Community Health Connection, Inc. CRS, Detroit, Michigan
  - McAuley Health Ctr. CRS, Grand Rapids, Michigan
  - Cooper Univ. Hosp. CRS, Camden, New Jersey
  - Cooper Hospital/Univ. Med. Ctr., The Cooper Early Intervention Program (EIP) CRS, Camden, New Jersey
  - New Jersey Medical School- Adult Clinical Research Ctr. CRS, Newark, New Jersey
  - South Jersey Infectious Disease, Cape Clinical Trials CRS, Somers Point, New Jersey
  - The Early Intervention Program at Kennedy Hosp. CRS, Voorhees Township, New Jersey
  - St. Vincent Hosp. & Med. Ctr. CRS, New York, New York
  - Bronx Prevention Center CRS, The Bronx, New York
  - Bronx-Lebanon Hosp. Ctr. CRS, The Bronx, New York
  - Montefiore Med. Ctr., AIDS Ctr. CRS, The Bronx, New York
  - PeaceHealth Med. Group - Hilyard Street Clinic CRS, Eugene, Oregon
  - Multnomah County Health Dept., HIV Health Services Ctr. CRS, Portland, Oregon
  - Legacy Clinic Good Samaritan CRS, Portland, Oregon
  - The Research & Education Group-Portland CRS, Portland, Oregon
  - Providence Portland Med. Ctr., Ambulatory Care and Education Ctr. CRS, Portland, Oregon
  - Kaiser Immune Deficiency Clinic of Portland CRS, Portland, Oregon
  - Legacy Clinic Emanuel CRS, Portland, Oregon
  - Oregon Health & Sciences Univ. Internal Medicine (L-475) CRS, Portland, Oregon
  - Philadelphia FIGHT - Dr. Jay Kostman CRS, Philadelphia, Pennsylvania
  - Temple Univ. School of Medicine CRS, Philadelphia, Pennsylvania
  - Albert Einstein Med. Ctr., Immunodeficiency Ctr. CRS, Philadelphia, Pennsylvania
  - MediCorp, Infectious Disease Associates CRS, Fredericksburg, Virginia
  - Hanover Med. Park (Mechanicsville, VA) CRS, Mechanicsville, Virginia
  - Eastern Virginia Med. School, Ctr. for the Comprehensive Care of Immune Deficiency CRS, Norfolk, Virginia
  - Petersburg Health Care Alliance CRS, Petersburg, Virginia
  - Vernon Harris East End Community Health Ctr. CRS, Richmond, Virginia
  - CrossOver Health Ctr. CRS, Richmond, Virginia
  - South Richmond Health Care Ctr. CRS, Richmond, Virginia
  - Hunter Holmes McGuire VAMC CRS, Richmond, Virginia
  - VCU Health Systems, Infectious Disease Clinic CRS, Richmond, Virginia

REFERENCES:
- [Background] Bunnell R, Ekwaru JP, Solberg P, Wamai N, Bikaako-Kajura W, Were W, Coutinho A, Liechty C, Madraa E, Rutherford G, Mermin J. Changes in sexual behavior and risk of HIV transmission after antiretroviral therapy and prevention interventions in rural Uganda. AIDS. 2006 Jan 2;20(1):85-92. doi: 10.1097/01.aids.0000196566.40702.28. PMID 16327323
- [Background] Kozal MJ, Amico KR, Chiarella J, Schreibman T, Cornman D, Fisher W, Fisher J, Friedland G. Antiretroviral resistance and high-risk transmission behavior among HIV-positive patients in clinical care. AIDS. 2004 Nov 5;18(16):2185-9. doi: 10.1097/00002030-200411050-00011. PMID 15577652
- [Background] Remien RH, Halkitis PN, O'Leary A, Wolitski RJ, Gomez CA. Risk Perception and sexual risk behaviors among HIV-positive men on antiretroviral therapy. AIDS Behav. 2005 Jun;9(2):167-76. doi: 10.1007/s10461-005-3898-7. PMID 15933836
- See also: Click here for more information on CPCRA 065 — http://clinicaltrials.gov/show/NCT00027352